CLINICAL TRIAL: NCT01619787
Title: Experimental Analysis of Price Changes and Food Purchases in Obese and Lean Mothers
Brief Title: Price Changes and Hypothetical Food Purchases in Adult Grocery Shoppers
Acronym: Grocery
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Epstein, SUNY Distinguished Professor of Pediatrics and Social and Preventive Medicine, State University of New York at Buffalo
Other Study IDs: 1090209-1-55244
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Effect of Taxes and Subsides on Food Purchases in Mothers

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the proposed study is to apply experimental economics in an online grocery store shopping model to examine the effects of pricing on hypothetical food purchases

DETAILED DESCRIPTION:
Participants will be lean and overweight primary grocery shoppers aged 18 years and older. Participants will be considered lean if their body mass index (BMI = kg/m2) is less than 29.9, overweight if their BMI is greater than or equal to 30.12 To meet eligibility for the study, participants must be the guardian of a child at least 2 years or older, do the primary grocery shopping for the family, they must also report being weekly household grocery shoppers, and purchase the majority of their household's groceries once a week.

ELIGIBILITY:
Inclusion Criteria:

18 or older primary shopper in the household, at least one child over 2 years of age

Exclusion Criteria:

eating disorders, not liking study foods

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lean and overweight Low and high socioeconimic status primary grocery shopper
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H Epstein, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Epstein LH, Paluch RA, Carr KA, Temple JL, Bickel WK, MacKillop J. Reinforcing value and hypothetical behavioral economic demand for food and their relation to BMI. Eat Behav. 2018 Apr;29:120-127. doi: 10.1016/j.eatbeh.2018.03.008. Epub 2018 Apr 3. PMID 29656049
- [Derived] Epstein LH, Finkelstein E, Raynor H, Nederkoorn C, Fletcher KD, Jankowiak N, Paluch RA. Experimental analysis of the effect of taxes and subsides on calories purchased in an on-line supermarket. Appetite. 2015 Dec;95:245-51. doi: 10.1016/j.appet.2015.06.020. Epub 2015 Jul 3. PMID 26145274
- [Derived] Epstein LH, Jankowiak N, Fletcher KD, Carr KA, Nederkoorn C, Raynor HA, Finkelstein E. Women who are motivated to eat and discount the future are more obese. Obesity (Silver Spring). 2014 Jun;22(6):1394-9. doi: 10.1002/oby.20661. Epub 2013 Dec 6. PMID 24311480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in the Western New York Area targeted primary household grocery shoppers through the local community during 2011-2013.
Pre-assignment Details: Interested eligible participants were screened and offered to start the study.
Groups:
- Online Grocery: All participants completed a baseline session where behavioral measures of delay discounting, relative reinforcing value and relative reinforcing efficacy were measured. Participants then completed five shopping sessions under various price conditions. Age and Body Mass Index were measured at the end of the six session study.
Period: Overall Study
Arm/Group | Online Grocery
Started | 217
Completed | 212
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Age and Body Mass Index (BMI) were measured at the end of the study; therefore 5 participants were lost to follow up and the baseline measures are reported on 212 participants.
Groups:
- Lean Participants: Participants whose baseline BMI is less than 25.
  All participants completed a baseline session where behavioral measures of delay discounting, relative reinforcing value and relative reinforcing efficacy were measured. Participants then completed five shopping sessions under various price conditions. Age and Body Mass Index were measured at the end of the six session study; therefore, 5 participants were lost to follow up and no age or body mass index are reported for these participants.
- Overweight/Obese Participants: Participants whose baseline BMI is greater than or equal to 25.
  All participants completed a baseline session where behavioral measures of delay discounting, relative reinforcing value and relative reinforcing efficacy were measured. Participants then completed five shopping sessions under various price conditions. Age and Body Mass Index were measured at the end of the six session study; therefore, 5 participants were lost to follow up and no age or body mass index are reported for these participants.
- Total: Total of all reporting groups
Arm/Group | Lean Participants | Overweight/Obese Participants | Total
Number analyzed (Participants) | 102 | 110 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (7.5) | 42.5 (7.4) | 42.7 (7.4)
Gender [Count of Participants; unit: Participants]
  Female | 99 | 105 | 204
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 100 | 110 | 210
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 22 | 36
  White | 79 | 83 | 162
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) was measured at the end of the sixth study session; therefore, 5 participants were lost to follow up and this is measured with 212 participants.
  kg/m^2 | 32.6 (6.6) | 22.2 (2.0) | 27.6 (7.2)
Relative Reinforcing Value High Energy Dense Foods (RRV HED) [Mean (Standard Deviation); unit: Highest Response schedule completed] — RRV was assessed using a computer program where subjects earned points toward food. Participants earned a point by clicking a mouse to meet schedule requirements, i.e. 20 clicks earned one portion of food on schedule one. Each subsequent schedule had double the requirements of the previous schedule. Participants were rewarded with their preferred food each time they completed the schedule requirements. The session ended when participants no longer wished to earn points towards food.
  Highest Response schedule completed | 13.8 (50.4) | 15.9 (25.1) | 14.7 (38.8)
Relative Reinforcing Value Low Energy Dense Foods (RRV LED) [Mean (Standard Deviation); unit: Highest response schedule completed] — RRV was assessed using a computer program where subjects earned points toward food. Participants earned a point by clicking a mouse to meet schedule requirements, i.e. 20 clicks earned one portion of food on schedule one. Each subsequent schedule had double the requirements of the previous schedule. Participants were rewarded with their preferred food each time they completed the schedule requirements. The session ended when participants no longer wished to earn points towards food.
  Highest response schedule completed | 26.0 (34.7) | 23.9 (30.4) | 25.2 (32.9)
Delay Discounting $10 reward (DD 10) [Mean (Standard Deviation); unit: indifference proportion*delay proportion] — The delay discounting task involved allowing participants to make choices between smaller immediate monetary rewards and a larger, fixed, delayed reward. Participants completed both increasing amount of the immediate reward, and decreasing amount of the immediate reward, in a randomized order, over a series of time delays (1 day, 2 days, etc). An indifference point was calculated as the amount of immediate reward that was equal to the delayed reward. From this area under the curve, or indifference proportion*delay proportion, was calculated, leading the a range of scores between 0 and 1.
  indifference proportion*delay proportion | 0.7 (0.3) | 0.6 (0.3) | 0.6 (0.3)
Delay Discounting $100 reward (DD 100) [Mean (Standard Deviation); unit: indifference proportion*delay proportion] — The delay discounting task involved allowing participants to make choices between smaller immediate monetary rewards and a larger, fixed, delayed reward. Participants completed both increasing amount of the immediate reward, and decreasing amount of the immediate reward, in a randomized order, over a series of time delays (1 day, 2 days, etc). An indifference point was calculated as the amount of immediate reward that was equal to the delayed reward. From this area under the curve, or indifference proportion*delay proportion, was calculated, leading the a range of scores between 0 and 1.
  indifference proportion*delay proportion | 0.7 (0.2) | 0.7 (0.3) | 0.7 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Energy Purchased as a Result of Taxes.
Description: Change in total calories as a result of taxes of 12.5% and 25%.
Time Frame: Study Completion
Population: Data is reported for 199 participants. Out of 217 participants who started the study, 5 participants were lost to follow up, 1 participant shopped in the same store twice, 2 participants had conditions that would affect shopping, 2 participants did not report minority status and 8 male participants were excluded due to the small sample number.
Measure: Least Squares Mean (Standard Error); unit: Total Calories Purchased
Groups:
- Lean Participants: Participants with BMI less than 25.
- Overweight/Obese Participants: Participants with BMI greater than or equal to 25.
Arm/Group | Online Grocery | Lean Participants | Overweight/Obese Participants
Number analyzed (Participants) | 199 | 97 | 102
Total Calories Purchased
  Calories Purchased in the Regular Condition | 10622.09 (329.04) | 10507.62 (427.92) | 10311.12 (456.04)
  Calories Purchased in the Tax 12.5 Condition | 10401.13 (292.12) | 10512.95 (523.10) | 9733.12 (385.34)
  Calories Purchased in the Tax 25 Condition | 10180.17 (304.13) | 10471.42 (464.73) | 10184.04 (436.78)

2. Primary Outcome: Change in Energy Purchased as a Result of Subsidies
Description: Change in total calories as a result of subsidies of 12.5% and 25%.
Time Frame: Study Completion
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Total Calories Purchased
Arm/Group | Online Grocery | Lean Participants | Overweight/Obese Participants
Number analyzed (Participants) | 199 | 97 | 102
Total Calories Purchased
  Calories Purchased in the Regular Condition | 10548.69 (316.69) | 10507.63 (437.92) | 10311.12 (456.04)
  Calories Purchased in the Subsidy 12.5 Condition | 10369.12 (283.95) | 10176.01 (442.21) | 9704.67 (405.05)
  Calories Purchased in the Subsidy 25 Condition | 10189.55 (300.85) | 11036.01 (519.23) | 10509.31 (426.99)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected at each of six study sessions scheduled one week apart.
Groups:
- Online Grocery: All participants completed a baseline session where behavioral measures of delay discounting, relative reinforcing value and relative reinforcing efficacy, along with the Three Factor Eating Questionnaire were measured. Participants then completed five shopping sessions under various price conditions. Age and Body Mass Index were measured at the end of the six session study.
Arm/Group | Online Grocery
Serious Adverse Events (participants affected / at risk) | 0/217
Other Adverse Events (participants affected / at risk) | 0/217

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No